CLINICAL TRIAL: NCT05023044
Title: Nonalcoholic Fatty Liver Disease In Persons Living With HIV Database Study
Brief Title: Nonalcoholic Fatty Liver Disease in HIV Database
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00316850; R01DK121378 (NIH)
Record Dates: First submitted 2021-08-06; First posted 2021-08-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: NAFLD; NASH - Nonalcoholic Steatohepatitis; Hiv
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fasting serum and plasma, DNA (in participants consenting to genetic research), PBMCs, stool, and snap frozen liver tissue will be banked in the NAFLD in HIV Database. Blood will be drawn for serum and plasma banking during screening and yearly visits on all participants enrolled in the study. If a standard of care liver biopsy is obtained at any time for any reason after the participant has signed the informed consent form, a portion of the liver sample will be collected for banking. The samples will be shipped on dry ice to the Indiana University Biorepository.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a spectrum of liver conditions associated with fat accumulation that ranges from benign, non-progressive liver fat accumulation to severe liver injury, cirrhosis, and liver failure. The spectrum of NAFLD encompasses simple nonalcoholic steatosis (nonalcoholic fatty liver [NAFL]) and nonalcoholic steatohepatitis (NASH) in which there is evidence of hepatocellular injury and/or fibrosis. NAFLD is the most common liver disease in adults and the second leading cause for liver transplantation in the U.S. The natural history of NAFLD in the general population has been well described. The NASH Clinical Research Network (NASH CRN) was established by the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) in 2002 to further the understanding of the diagnosis, mechanisms, progression and therapies of NASH. This effort has resulted in numerous seminal studies in the field. However, NASH CRN studies have systematically excluded persons living with HIV (PLWH) , as NAFLD in PLWH was thought to be different from that in the general population due to HIV infection, antiretroviral therapy (ART), concomitant medications and co-infections. This resulted in major knowledge gaps regarding NAFLD in the setting of HIV infection. Thus, the natural history of NAFLD in PLWH is largely unknown. The goal of this ancillary study of NAFLD and NASH in Adults with HIV (HIV NASH CRN), is to conduct a prospective, observational, multicenter study of NAFLD in PLWH (HIV-associated NAFLD).

DETAILED DESCRIPTION:
NAFLD is the most prevalent of all liver disorders and is the most common cause of chronic aminotransferase elevations in the U.S. With the availability of highly effective ART, chronic liver disease has become a leading cause of non-AIDS related morbidity and mortality in PLWH. NAFLD is projected to become the leading cause of liver disease in the aging HIV population. While there is evidence that both Hepatitis B and Hepatitis C infection follow an accelerated course in PLWH, it is unknown if NAFLD is also accelerated in PLWH. Unlike NAFLD in the general population, there is a significant lack of characterization of the natural history of NAFLD in PLWH. This prospective observational study of PLWH with NAFLD will examine the natural history of HIV-associated NAFLD. It will also test the accuracy of non-invasive assessments of advanced fibrosis in detecting histologically confirmed advanced fibrosis in PLWH, and establish a robust biospecimen bank (plasma, serum, genomic DNA, and urine; peripheral blood mononuclear cells (PBMCs) and stool at select sites).

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* ≥18 of age at time of initial screening
* HIV suppression with HIV RNA <200 copies/ml on stable ART for ≥ 6 months and no change in ART class for ≥ 3 months, prior to enrollment
* Participants must meet at least one of the following inclusion criteria:

  * Histologically confirmed NAFLD [defined as NAFL (>5% steatosis, with or without lobular or portal inflammation), borderline NASH or definitive NASH] within 6 months prior to screening (per local pathology report)
  * Liver stiffness measurement (LSM) ≥6 kPa from FibroScan exam performed during screening or within 12 months prior to screening and a diagnosis of NAFLD based on clinical and imaging (FibroScan CAP≥263 dB/m, ultrasound, CT or MRI) diagnosis at any time
  * LSM ≥8 kPa from FibroScan exam performed during screening or within 12 months prior to screening, in the absence of CAP ≥263 dB/m
* Able to provide written informed consent to part
* Willingness to be in the study for 1 or more years
* Provision of written informed consent

Exclusion Criteria:

* Positive hepatitis B surface antigen
* Evidence of recent or current hepatitis C virus (HCV) as marked by the presence of anti-HCV antibody with detectable HCV RNA in serum within 3 years prior to enrollment. Participants with anti-HCV antibody positivity who have undetectable HCV RNA 3 years prior to enrollment (either due to spontaneous clearance or clearance with treatment) will be eligible to participate if HCV RNA at entry remains undetected
* Significant alcohol consumption (≥ 3 drinks daily on average in men and ≥ 2 drinks daily on average in women)
* Evidence of other causes of chronic liver disease
* History of prolonged (> 1 month) total parenteral nutrition within a 6-month period before liver biopsy or before baseline FibroScan VCTE exam
* Short bowel syndrome
* History of biliopancreatic diversion
* History of bariatric surgery within 2 years of enrollment (participants expecting to undergo bariatric surgery can be enrolled prior to the procedure)
* Solid organ transplant recipients
* Other condition that is likely to interfere with study follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 participants who are PLWH at least 18 years of age with a diagnosis of NAFLD, NASH, or NASH-related cirrhosis, supported by either a recent liver biopsy or clinical and imaging criteria
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2031-09-01 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in liver stiffness measurement (LSM) measured by VCTE from baseline to one year | Baseline and 1 year
  Vibration-controlled transient elastography (VCTE) measures the speed of a mechanically generated shear wave across the liver to derive a liver stiffness measurement (LSM), which corresponds to the liver fibrosis stage. LSM is measured in kilopascals (kPa).
Change in controlled attenuation parameter (CAP) measured by VCTE from baseline to one year | Baseline and 1 year
  Controlled attenuation parameter (CAP) measures the increased attenuation of ultrasound waves when traveling through fat in the liver and is a non-invasive method to assess hepatic steatosis. CAP is measured in decibels per meter (dB/m).

CONTACTS AND LOCATIONS:
Overall Officials: Tinsay A Woreta, MD, MPH, Principal Investigator — Johns Hopkins University; Samer Gawrieh, MD, Principal Investigator — Indiana University
Locations (8):
- United States (8):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University, Durham, North Carolina
  - University of Texas, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joshi D, O'Grady J, Dieterich D, Gazzard B, Agarwal K. Increasing burden of liver disease in patients with HIV infection. Lancet. 2011 Apr 2;377(9772):1198-209. doi: 10.1016/S0140-6736(10)62001-6. PMID 21459211
- [Background] Price JC, Thio CL. Liver disease in the HIV-infected individual. Clin Gastroenterol Hepatol. 2010 Dec;8(12):1002-12. doi: 10.1016/j.cgh.2010.08.024. Epub 2010 Sep 17. PMID 20851211
- [Background] Smith CJ, Ryom L, Weber R, Morlat P, Pradier C, Reiss P, Kowalska JD, de Wit S, Law M, el Sadr W, Kirk O, Friis-Moller N, Monforte Ad, Phillips AN, Sabin CA, Lundgren JD; D:A:D Study Group. Trends in underlying causes of death in people with HIV from 1999 to 2011 (D:A:D): a multicohort collaboration. Lancet. 2014 Jul 19;384(9939):241-8. doi: 10.1016/S0140-6736(14)60604-8. PMID 25042234
- [Background] Crum-Cianflone NF. Editorial Commentary: Elevated Aminotransferase Levels Among HIV-Infected Persons: What's Lurking Under the Surface? Clin Infect Dis. 2015 May 15;60(10):1579-81. doi: 10.1093/cid/civ106. Epub 2015 Feb 13. No abstract available. PMID 25681377
- [Background] Crum-Cianflone N, Dilay A, Collins G, Asher D, Campin R, Medina S, Goodman Z, Parker R, Lifson A, Capozza T, Bavaro M, Hale B, Hames C. Nonalcoholic fatty liver disease among HIV-infected persons. J Acquir Immune Defic Syndr. 2009 Apr 15;50(5):464-73. doi: 10.1097/QAI.0b013e318198a88a. PMID 19225402
- [Background] Siddiqui MS, Vuppalanchi R, Van Natta ML, Hallinan E, Kowdley KV, Abdelmalek M, Neuschwander-Tetri BA, Loomba R, Dasarathy S, Brandman D, Doo E, Tonascia JA, Kleiner DE, Chalasani N, Sanyal AJ; NASH Clinical Research Network. Vibration-Controlled Transient Elastography to Assess Fibrosis and Steatosis in Patients With Nonalcoholic Fatty Liver Disease. Clin Gastroenterol Hepatol. 2019 Jan;17(1):156-163.e2. doi: 10.1016/j.cgh.2018.04.043. Epub 2018 Apr 26. PMID 29705261
- [Background] Sterling RK, Smith PG, Brunt EM. Hepatic steatosis in human immunodeficiency virus: a prospective study in patients without viral hepatitis, diabetes, or alcohol abuse. J Clin Gastroenterol. 2013 Feb;47(2):182-7. doi: 10.1097/MCG.0b013e318264181d. PMID 23059409
- [Background] Vilar-Gomez E, Chalasani N. Non-invasive assessment of non-alcoholic fatty liver disease: Clinical prediction rules and blood-based biomarkers. J Hepatol. 2018 Feb;68(2):305-315. doi: 10.1016/j.jhep.2017.11.013. Epub 2017 Dec 2. PMID 29154965